CLINICAL TRIAL: NCT04214977
Title: Spinal Anesthesia Versus General Anesthesia Using Laryngeal Mask Airway for Anorectal Surgeries in Prone Position: A Controlled Clinical Trial
Brief Title: Spinal Anesthesia Versus General Anesthesia Using Laryngeal Mask Airway for Anorectal Surgeries in Prone Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Mahmoud M. Almustafa, Principal Investigator, University of Jordan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 67/2019/1174
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia; Anorectal Surgery
Keywords: Anorectal surgeries; prone; spinal anaesthesia; general anaesthesia; laryngeal mask
MeSH Terms: interventions — Anesthesia, Spinal; Prone Position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group S (Experimental): Patients in group S had spinal anesthesia in the sitting position under complete aseptic technique through a standard mid-line approach. The patient was then asked to turn him- or herself into the prone position on the surgical table with the help of the surgical and anesthetic teams.
  Interventions: Procedure: Spinal Anesthesia for Anorectal Surgeries in Prone Position
- group L (Experimental): Patients in group L received standard general anesthesia. Proper (weight-based) classic laryngeal mask airway was then blindly inserted.
  Interventions: Procedure: General Anesthesia Using Laryngeal Mask Airway for Anorectal Surgeries in Prone Position

INTERVENTIONS:
Procedure: Spinal Anesthesia for Anorectal Surgeries in Prone Position — Spinal anesthesia in sitting position was done under complete aseptic technique through a standard midline approach. One and a half millilitres of 0.5% bupivacaine (7.5 mg) was injected through a 25 Gauge pencil-point needle into the subarachnoid space at L3-L4 or L4-L5 interspace. All patients were kept in a head-up position for 3 minutes. The patient was then asked to turn him- or herself into the prone position on the surgical table with the help of the surgical and anesthetic teams.
  Arms: group S
Procedure: General Anesthesia Using Laryngeal Mask Airway for Anorectal Surgeries in Prone Position — General anesthesia was induced using fentanyl 2 mcg/kg and Propofol 2-3 mg/kg. Any stomach contents were then suctioned through an oro-gastric tube to reduce the risk of regurgitation. Proper (weight-based) classic laryngeal mask airway was then blindly inserted. laryngeal mask airway was then properly fixed to the face and anesthesia was maintained with isoflurane 1-2% in 50% Oxygen/air mixture.
  Arms: group L

SUMMARY:
Anorectal surgeries are of the commonest elective surgeries that are performed worldwide under different types of anaesthesia. The aim of this prospective interventional study was to compare the use of general anaesthesia (GA) using a laryngeal mask airway (LMA) with spinal anesthesia (SA) in anorectal surgeries.

DETAILED DESCRIPTION:
Anorectal surgeries are of the most frequently performed procedures worldwide. These procedures are commonly performed in prone position as it offers sufficient exposure and provides enough surgical space. Choosing the suitable anesthetic technique will help in reducing perioperative complications in patients undergoing surgical procedures in prone position, by taking into consideration changes in cardiovascular and pulmonary physiology, airway management, and proper positioning for the prevention of direct and indirect pressure injuries. The aim of this prospective interventional controlled study was to compare the use of general anesthesia (GA) using a laryngeal mask airway (LMA) with spinal anesthesia (SA) in anorectal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective anorectal surgery (perianal fistula surgery, haemorrhoidectomy, perianal abscess, pilonidal sinus, anal fissure or evaluation under anaesthesia).
* patients older than 16-years old.
* patients who have ASA score I-III.
* Patients whose BMI is less than 35 kg/m2.

Exclusion Criteria:

* any patient who refused to participate in the study.
* patients with surgeries for anal or rectal tumors.
* any patient with expected surgery's duration more than 90 minutes
* patients with uncontrolled respiratory conditions
* any patient whose preoperative assessment was suggestive of possibility of difficult airway.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
comparison was between the induction and emergence anesthesia times needed in each technique | 4 months
  In this group (L) the investigators defined induction time (T1) as the time from completion of initial monitoring until the patient is positioned prone. Emergence time (T2) was defined as the time from the end of surgical dressing till the removal of LMA in the supine position and the patient is ready for transfer to PACU.
  . In this group the investigators defined induction time (T1) as the time from the end of initial monitoring till the patient is positioned in prone position, and (T2) as the time from the end of surgical dressing till the patient is turned to supine position on the bed and ready to be transferred to PACU.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No